CLINICAL TRIAL: NCT02125942
Title: Pilot Study of Central Meditation and Imagery Therapy for Borderline Personality Disorder
Brief Title: Central Meditation and Imagery Therapy for Augmentation of Borderline Personality Disorder Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMIT1044
Record Dates: First submitted 2014-04-26; First posted 2014-04-29 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- meditation (Experimental): Central Meditation and Imagery Therapy
  Interventions: Behavioral: Central Meditation and Imagery Therapy
- wait list (No Intervention): waiting list

INTERVENTIONS:
Behavioral: Central Meditation and Imagery Therapy — mindfulness, guided imagery, meditation
  Arms: meditation

SUMMARY:
Borderline personality disorder is a severe psychiatric disorder marked by emotional instability, difficulty with interpersonal relationships, and self-harming behaviors. Despite receiving psychotherapy for borderline personality disorder, studies show that patient recovery is slow, and there is a high rate of self injury and suicide attempts early in treatment. There is thus a clear need to provide therapies to augment psychotherapy. We will conduct a pilot trial to determine whether a 6-week Central Meditation and Imagery Therapy (CMIT) is feasible for subjects with borderline personality disorder to undergo when added on to psychotherapy treatment. CMIT is a non-validated therapy that combines principles of mindfulness with meditation techniques and guided imagery. Sessions led by a trained clinician in a group setting once a week, and participants are asked to complete daily home practice.

The trial will involve 16 participants, all currently undergoing psychotherapy for borderline personality disorder. Participants will be randomly assigned to either a CMIT group that lasts 6 weeks, or a wait list group. Those in the wait list group will be able to receive CMIT after 6 weeks. All participants will continue to receive psychotherapy throughout the trial.

During the trial, we will also obtain preliminary data to help understand whether CMIT may result in psychological benefits for participants. This will include measuring the pulse in order to determine variation in beat to beat intervals of the heart during psychological tests, and filling out questionnaires before and after participation in CMIT.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic criteria for BPD according to DSM-IV criteria
* Meeting the diagnostic criteria for BPD based on the Diagnostic Interview for Borderline - Revised
* Currently receiving psychotherapy.
* English language proficiency to understand written and oral communication

Exclusion Criteria:

* Active suicidality or suicidal intent as identified on the Columbia Suicide Severity Rating Scale
* Suicide attempt within the past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Borderline Symptoms | 6 weeks
  Borderline Symptom List

SECONDARY OUTCOMES:
Depression | 6 weeks
  Quick Inventory of Depressive Symptoms
Anxiety | 6 weeks
  Trait Anxiety Inventory
Positive Affect | 6 weeks
  Positive and Negative Affect Scale

OTHER OUTCOMES:
Heart rate variability | 6 weeks
  Resting heart rate variability

CONTACTS AND LOCATIONS:
Overall Officials: Felipe A Jain, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793